CLINICAL TRIAL: NCT03981120
Title: The Effect of Acupuncture on in Vitro Fertilization Outcomes in Women Undergoing Euploid Embryo Transfer - A Pilot Study
Brief Title: The Effect of Acupuncture on Pregnancy Rates in Women Undergoing in Vitro Fertilization With Preimplantation Genetic Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Gary Nakhuda, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Acupuncture and IVF
Record Dates: First submitted 2019-05-30; First posted 2019-06-10 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Infertility; Aneuploidy
Keywords: In-vitro fertilization; acupuncture; preimplantation genetic screening; pregnancy; laser; miscarriage
MeSH Terms: conditions — Infertility; Aneuploidy; Abortion, Spontaneous | interventions — Lasers

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be assigned a computer generated code to be used on data collection forms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Group (No Intervention): Patients in the control arm will not undergo laser and acupuncture treatment. The treatment and control group will be compared to the baseline pregnancy rate of women meeting the same inclusion and exclusion criteria from the clinic through a chart review over the two years prior to initiation of the study.
- Laser and Acupuncture Group (Experimental): The patients in the treatment arm will have 7 treatments before transfer (2-4 sessions a week), for the 3 weeks from starting estrace leading to the day before embryo transfer, then one (before and after transfer) on the day of transfer (total 8 sessions). Each treatment leading up to transfer day treatment consists of:
  1. Traditional Acupuncture at points Sp9 to SP6 EA2Hz Milliamp (Pantheon device), ST-36 B, LI4 unilateral, LV3 unilateral and/or LU7 unilateral, K6 unilateral.
  2. Bioflex Array (Photobiomodulation) - simultaneously array placements with each treatment over the sacrum (points BL-31, BL 32, BL 33 BL 34, DU2, DU3) and lower Abdomen above uterus (Ren 2 to Ren 6)
  3. Laser acupuncture over ST-9, ST10, SJ 17, ST-11. Ren 3 and Ren 4. 6.75 J per point at ST 9, ST10 (over carotid) and SJ17 (vertebral artery).
  On the day of FET on site at IVF clinic there will be a before and after traditional and laser acupuncture treatment.
  Interventions: Procedure: Laser and Traditional Acupuncture

INTERVENTIONS:
Procedure: Laser and Traditional Acupuncture — Acupuncture (traditional and laser) and photobiomodulation will be performed by a certified acupuncturist on-site with experience in reproductive health and the initial visit will include an assessment and traditional Chinese medicine (TCM) diagnosis.
  Arms: Laser and Acupuncture Group

SUMMARY:
While IVF offers an effective treatment for infertility, a significant proportion of IVF cycles still result in failed implantation and early miscarriage. As such, new therapies that improve pregnancy outcomes are highly desirable. Both traditional and laser acupuncture during the IVF cycle has become a popular option for women looking to improve their pregnancy rates. However, studies looking to understand the effects of acupuncture on IVF have demonstrated contradicting results. While some studies show an improvement in pregnancy rates in women undergoing IVF with traditional acupuncture treatment, other studies show no difference. Moreover, there are few studies exploring the role of laser and traditional acupuncture in IVF cycles and the studies done thus far have shown no change in pregnancy rates. However, there have been no studies to-date that have looked at women who are receiving IVF for embryos with normal genetics. This is important because embryos with abnormal genetics are a major reason for failed implantation and miscarriage, which can make the effects of acupuncture on pregnancy rates difficult to evaluate. This study is a pilot study looking to better understand the role of laser and traditional acupuncture as a supplemental treatment in women undergoing euploid (normal genetics) embryo transfer. This is the first study to include only genetically normal embryos, which may help to better understand the effects of laser and traditional acupuncture on IVF outcomes.

DETAILED DESCRIPTION:
Purpose:

To assess the feasibility and preliminary outcomes of a single-blinded randomized clinical trial evaluating the effect of laser and traditional acupuncture during the IVF cycle on pregnancy outcomes in women undergoing euploid embryo transfer.

Hypothesis:

A single-blinded randomized clinical trial evaluating the effects and reproductive outcomes of laser and traditional acupuncture during the IVF cycle will be acceptable to patients and feasible for a large fertility clinic.

Justification:

IVF is a costly treatment option for women, their partners, and the public. Therefore, new therapies that improve reproductive and health outcomes are highly desirable. Furthermore, the economic burden of IVF is directly related to the number of attempted cycles, and hence there is a growing interest in the use of adjuvant therapies to optimize pregnancy outcomes on a per cycle basis.

Acupuncture, both traditional and laser, has become a popular adjuvant therapy for women undergoing IVF treatment. Previous studies attempting to validate the effects of traditional acupuncture on IVF outcomes have demonstrated contradicting results. Importantly, none of the prior studies controlled for the effect of embryonic aneuploidy, which is a major contributor to implantation failure and early miscarriage. Further, there are very few studies assessing the effects of laser and traditional acupuncture on IVF outcomes and no studies to date that take into account embryo genetics.

Hence, the purpose of this study is to investigate the feasibility of a randomized clinical trial assessing the effects of laser and traditional acupuncture on IVF outcomes in women undergoing euploid embryo transfer after complete chromosomal screening, thereby controlling for a normal karyotype and allowing for a more meaningful analysis of the effect of laser and traditional acupuncture on IVF outcomes.

Objectives:

1. To assess patient acceptance and clinical feasibility of a well-designed randomized clinical pilot study comparing the effects of a clinical-dose (8 total sessions) of laser and needle acupuncture on pregnancy outcomes in IVF.
2. To generate preliminary results based on a feasible study design that may inform the implementation of a larger randomized clinical study in the future.

Research design:

One hundred patients undergoing IVF with preimplantation genetics screening will be randomized using a computer-generated block randomization method to either the laser and traditional acupuncture (n = 50) or standard-of-care (n = 50) arm. The laser acupuncture arm will be offered treatment 3 times a week starting from menses, plus an additional treatment before embryo transfer (ET). The goal is to have completed 7 treatments prior to ET, for a total of 8 treatments (last treatment done at Olive Centre right before ET). Patients in the standard-of-care arm will receive standard treatment. Physicians and nurses will be blinded to the groups assigned and will provide the same standard of care to both groups. Participants will be asked to complete a short survey following each laser acupuncture treatment.

Study procedure:

Participants in the laser and needle acupuncture arm will be offered treatment 2-4 times a week starting from menses, plus an additional treatment before ET. The goal is to have completed 7 treatments prior to ET, then one one on the day of ET (before and after transfer), for a total of 8 treatment sessions. Participants will be asked to complete a short survey following each laser and traditional acupuncture session.

Because the results of the preimplantation genetic screening (PGS) do not return with enough time for a fresh embryo transfer, all PGS embryos are transferred as part of a frozen ET. Unfortunately, there are no consensus protocols on the use of acupuncture in either frozen or fresh embryo IVF transfers. As such, we have used the expert opinions of several registered acupuncturists skilled in reproductive health to arrive at a consensus laser acupuncture protocol that is appropriate for a frozen-embryo transfer. Full details of the protocol are included in the Research Proposal.

Laser and traditional acupuncture will be performed by a certified acupuncturist skilled in reproductive health and experienced with use of laser and needle acupuncture in IVF. Physicians and nurses will be blinded to the groups assigned. The following certified acupuncturists will be performing the acupunctures:

Lorne Brown Ryan Funk Emilie Salomons Christina Ceconni Allison Locke Kathleen Lee Bronwyn Melville There are fewer variables with laser acupuncture than traditional acupuncture. The amount of energy and distance from each acupoint are the same, so there is less variation between providers. With traditional acupuncture, there is difference in needle depth of penetration, pressure, etc. Additionally, while it would be ideal for the same acupuncturist to provide all the treatment, this isn't feasible for the acupuncture clinic.

The reference arm will receive standard treatment.

The questionnaire surveys will be given to the patient participants after each laser acupuncture session if they are in the acupuncture group, and after their embryo transfer if they are from the standard care group. The study participants will be taken to a different room/office within the clinic to complete the surveys. To ensure blinding, the questionnaires will be provided by research staff not involved in the direct care of the patients. After completing the survey, the participant will place it in a sealed envelope.

This way, the participant responses are anonymized, with only the participant identification number on the forms, and no other patient-identifying information. The responses will not be made known to the physicians and nurses.

Statistical analysis:

Feasibility outcomes to be assessed include recruitment rate, refusal rate, retention rate, non-compliance rate, ability to maintain blindedness of healthcare staff, inclusion of all important data points, and determination of centre willingness and capacity.

Success of feasibility will be determined by the following criteria:

* At least 70% of all eligible participants choose to participate
* At least 90% retention of those that choose to participate
* At least 90% of all recruited participants complete six acupuncture sessions and the follow up survey
* At least 95% maintained blindedness of healthcare providers

ELIGIBILITY:
Inclusion Criteria:

* use of preimplantation genetic screening
* treatment with IVF/intracytoplasmatic sperm injection (ICSI)
* age <40
* BMI <35

Exclusion Criteria:

* three or more prior failed IVF cycles with euploid embryo transfer
* known structural or anatomic causes of infertility
* male factor infertility
* patients already receiving concomitant treatment within the last 3 months (e.g. reflexology, acupuncture, herbal supplements, meditation).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Pregnancy Rate | From date of embryo transfer until the date of first documented pregnancy, whichever comes first, up to 12 months
  Pregnancy beyond 10 weeks' gestation

SECONDARY OUTCOMES:
Biochemical Pregnancy Rate | From date of embryo transfer until the date of first documented biochemical pregnancy, whichever comes first, up to 12 months
  positive human chorionic gonadotropin (hCG) serum or urine test > or = 11 days after embryo transfer
Cumulative Pregnancy Rate | From date of embryo transfer until the date of first documented intrauterine pregnancy, whichever comes first, up to 12 months
  Presence of at least one intrauterine gestational sac or fetal heartbeat confirmed by ultrasound 4-6 weeks after embryo transfer
Live Birth Rate | From date of embryo transfer until the date of birth, whichever comes first, up to 12 months
  Baby born alive after 24 weeks gestation

OTHER OUTCOMES:
Rate of miscarriage | From date of embryo transfer until diagnosis, up to 12 months.
  Loss of pregnancy
Rate of adverse events | Any time during study period up to 12 months
  Any unfavourable outcome from medication or procedures.

IPD SHARING:
Plan to Share IPD: Yes
The de-identified research data will be deposited into a publicly accessible database after publication. This data includes demographics, treatment protocols, pregnancy outcomes, and other research-related information. At no time will identifying information, such their names, birth dates or street addresses be included in such data.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available within 6 months after the completion of the study.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will need to sign a Data Access Agreement

REFERENCES:
- [Background] Manheimer E. Selecting a control for in vitro fertilization and acupuncture randomized controlled trials (RCTs): how sham controls may unnecessarily complicate the RCT evidence base. Fertil Steril. 2011 Jun 30;95(8):2456-61. doi: 10.1016/j.fertnstert.2011.04.040. Epub 2011 May 13. PMID 21570069
- [Background] Zheng CH, Huang GY, Zhang MM, Wang W. Effects of acupuncture on pregnancy rates in women undergoing in vitro fertilization: a systematic review and meta-analysis. Fertil Steril. 2012 Mar;97(3):599-611. doi: 10.1016/j.fertnstert.2011.12.007. Epub 2012 Jan 11. PMID 22243605
- [Background] Zhang Y, Phy J, Scott-Johnson C, Garos S, Orlando J, Prien S, Huang JC. Effects of a Delphi consensus acupuncture treatment protocol on the levels of stress and vascular tone in women undergoing in-vitro fertilization: a randomized clinical trial protocol. BMC Complement Altern Med. 2017 Apr 4;17(1):197. doi: 10.1186/s12906-017-1693-4. PMID 28376836
- [Background] Shen C, Wu M, Shu D, Zhao X, Gao Y. The role of acupuncture in in vitro fertilization: a systematic review and meta-analysis. Gynecol Obstet Invest. 2015;79(1):1-12. doi: 10.1159/000362231. Epub 2014 May 16. PMID 24854767
- [Background] Qian Y, Xia XR, Ochin H, Huang C, Gao C, Gao L, Cui YG, Liu JY, Meng Y. Therapeutic effect of acupuncture on the outcomes of in vitro fertilization: a systematic review and meta-analysis. Arch Gynecol Obstet. 2017 Mar;295(3):543-558. doi: 10.1007/s00404-016-4255-y. Epub 2016 Dec 19. PMID 27995371
- [Background] Manheimer E, Zhang G, Udoff L, Haramati A, Langenberg P, Berman BM, Bouter LM. Effects of acupuncture on rates of pregnancy and live birth among women undergoing in vitro fertilisation: systematic review and meta-analysis. BMJ. 2008 Mar 8;336(7643):545-9. doi: 10.1136/bmj.39471.430451.BE. Epub 2008 Feb 7. PMID 18258932
- [Background] Cheong YC, Dix S, Hung Yu Ng E, Ledger WL, Farquhar C. Acupuncture and assisted reproductive technology. Cochrane Database Syst Rev. 2013 Jul 26;2013(7):CD006920. doi: 10.1002/14651858.CD006920.pub3. PMID 23888428
- [Background] El-Toukhy T, Khalaf Y. The impact of acupuncture on assisted reproductive technology outcome. Curr Opin Obstet Gynecol. 2009 Jun;21(3):240-6. doi: 10.1097/GCO.0b013e3283292491. PMID 19276803
- [Background] El-Toukhy T, Sunkara SK, Khairy M, Dyer R, Khalaf Y, Coomarasamy A. A systematic review and meta-analysis of acupuncture in in vitro fertilisation. BJOG. 2008 Sep;115(10):1203-13. doi: 10.1111/j.1471-0528.2008.01838.x. Epub 2008 Jul 23. PMID 18652588
- [Background] Manheimer E, van der Windt D, Cheng K, Stafford K, Liu J, Tierney J, Lao L, Berman BM, Langenberg P, Bouter LM. The effects of acupuncture on rates of clinical pregnancy among women undergoing in vitro fertilization: a systematic review and meta-analysis. Hum Reprod Update. 2013 Nov-Dec;19(6):696-713. doi: 10.1093/humupd/dmt026. Epub 2013 Jun 27. PMID 23814102
- [Background] Kung A, Munne S, Bankowski B, Coates A, Wells D. Validation of next-generation sequencing for comprehensive chromosome screening of embryos. Reprod Biomed Online. 2015 Dec;31(6):760-9. doi: 10.1016/j.rbmo.2015.09.002. Epub 2015 Sep 9. PMID 26520420
- [Background] Deng S, Zhao X, DU R, He SI, Wen Y, Huang L, Tian G, Zhang C, Meng Z, Shi X. Is acupuncture no more than a placebo? Extensive discussion required about possible bias. Exp Ther Med. 2015 Oct;10(4):1247-1252. doi: 10.3892/etm.2015.2653. Epub 2015 Jul 23. PMID 26622473
- [Background] Anderson B, Rosenthal L. Acupuncture and in vitro fertilization: critique of the evidence and application to clinical practice. Complement Ther Clin Pract. 2013 Feb;19(1):1-5. doi: 10.1016/j.ctcp.2012.11.002. Epub 2012 Dec 14. PMID 23337556
- [Background] Smith CA, Grant S, Lyttleton J, Cochrane S. Using a Delphi consensus process to develop an acupuncture treatment protocol by consensus for women undergoing Assisted Reproductive Technology (ART) treatment. BMC Complement Altern Med. 2012 Jul 7;12:88. doi: 10.1186/1472-6882-12-88. PMID 22769059
- [Background] Smith CA, de Lacey S, Chapman M, Ratcliffe J, Norman RJ, Johnson N, Sacks G, Lyttleton J, Boothroyd C. Acupuncture to improve live birth rates for women undergoing in vitro fertilization: a protocol for a randomized controlled trial. Trials. 2012 May 18;13:60. doi: 10.1186/1745-6215-13-60. PMID 22607192
- [Background] Nandi A, Shah A, Gudi A, Homburg R. Acupuncture in IVF: A review of current literature. J Obstet Gynaecol. 2014 Oct;34(7):555-61. doi: 10.3109/01443615.2014.919997. Epub 2014 Jun 9. PMID 24911326
- [Background] So EW, Ng EH, Wong YY, Lau EY, Yeung WS, Ho PC. A randomized double blind comparison of real and placebo acupuncture in IVF treatment. Hum Reprod. 2009 Feb;24(2):341-8. doi: 10.1093/humrep/den380. Epub 2008 Oct 21. PMID 18940896
- [Background] Dickersin K, Manheimer E. The Cochrane Collaboration: evaluation of health care and services using systematic reviews of the results of randomized controlled trials. Clin Obstet Gynecol. 1998 Jun;41(2):315-31. doi: 10.1097/00003081-199806000-00012. No abstract available. PMID 9646964
- [Background] Kaptchuk TJ, Stason WB, Davis RB, Legedza AR, Schnyer RN, Kerr CE, Stone DA, Nam BH, Kirsch I, Goldman RH. Sham device v inert pill: randomised controlled trial of two placebo treatments. BMJ. 2006 Feb 18;332(7538):391-7. doi: 10.1136/bmj.38726.603310.55. Epub 2006 Feb 1. PMID 16452103